CLINICAL TRIAL: NCT06726135
Title: The National Rehabilitation Centre Dataset. Development of a Minimum Dataset for Multidisciplinary Rehabilitation: a Modified E-Delphi Study
Brief Title: The NRC Dataset. Developing a Minimum Dataset for Multidisciplinary Rehabilitation: a Modified E-Delphi Study
Status: Not yet recruiting | Type: Observational
Sponsor: ThomasCorbett (Other)
Collaborators: Nottingham University Hospital NHS Trust (Unknown)
Responsible Party: Sponsor-Investigator, ThomasCorbett, Chief Investigator, Nottingham University Hospitals NHS Trust
Organization: Nottingham University Hospitals NHS Trust (Other)
Other Study IDs: 345539
Record Dates: First submitted 2024-12-05; First posted 2024-12-10 (Actual); Last update posted 2024-12-19 (Actual); Status verified 2024-12

CONDITIONS: Pain; Traumatic Brain Injury; Major Trauma; Multiple Sclerosis; Amputees / Rehabilitation; Spinal Cord Injuries (SCI); Functional Neurological Disorder; Intensive Care Unit (ICU) Acquired Weakness (ICU - AW); Trauma Related Injuries
Keywords: E-delphi; Delphi; Multidisciplinary; Rehabilitation; Core outcome set; Dataset; national rehabilitation centre; outcome measure instruments; inpatient
MeSH Terms: conditions — Pain; Brain Injuries, Traumatic; Multiple Sclerosis; Spinal Cord Injuries; Conversion Disorder

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Experts in the field of rehabilitation with knowledge in outcome monitoring and service evaluation: This study has one study cohort, consisting of a diverse panel of expert clinicians, researchers and managers from a variety of professional backgrounds.
  These study participants will be purposefully selected based on their knowledge of which demographic, socio-economic and healthcare related variables, as well as any associated outcome measure instruments should be collected as part of a rehabilitation dataset to evaluate the clinical efficacy and cost effectiveness of inpatient multidisciplinary rehabilitation.

SUMMARY:
Several rehabilitation datasets are presently in use for specific patient groups in England. The 'National Clinical Audit of Specialist Rehabilitation for patients with complex needs following major injury' (NCASRI) evaluated outcomes within a cohort of Major Trauma patients between 2015 and 2018 using data from two of these datasets. The NCASRI project outlined some of the shortcomings of the pre-existing datasets and highlighted the need for a single National Rehabilitation Dataset to provide long term evaluation of a variety of patient presentations.

The proposed study will seek to develop such a dataset by means of an E-delphi study. This study will seek consensus from a panel of experts on the data items required to measure the effectiveness and socio-economic impact of multidisciplinary inpatient rehabilitation. Providing commissioners, researchers and clinicians with the data required to improve patient care, conduct research and develop rehabilitation services.

There are three potential phases to this study:

* Phase one involves the establishment of a core domain set, outlining what information (data) should be included in the NRC core dataset.
* Phase one will consist of at least 2 rounds of voting, with successive rounds of voting undertaken until an a-priori consensus of 70% is reached for all core data items marked as mandatory/critical data in fitting OMERACT guidelines.
* After 2 rounds, any data item that have reached consensus will be included in the final dataset. These core domain (data items) will then be excluded from subsequent rounds of voting.
* A maximum of 4 rounds will be allowed in Phase 1. At which point the highest-ranking data items remaining with a consensus above 60% from each of the pre-identified categories will be included in the final dataset.
* Phase two will explore what tools should be used to collect the core domains (outcome measure instruments) for each category outlined in phase 1.
* Phase 2 will follow the same protocol for including outcome measure instruments into the core outcome set as were required to include core data items from phase 1.
* If a consensus of equal or greater than 60% cannot be reached using an E-Delphi method in either phase 1 or phase 2 then a virtual meeting will be held amongst all expert panel members to reach consensus using a nominal group technique (phase 3).

DETAILED DESCRIPTION:
This methodology of this modified e-Delphi study has been informed by guidelines on 'how to develop core domain/outcome sets' and 'how to conduct Delphi studies' by the Initiative on Methods, Measurements and Pain Assessment in Clinical Trials (IMMPACT), the Core Outcome Measures in Effectiveness Trials (COMET) group, the Outcome Measures in Rheumatology (OMERACT) group and The Consensus-based Standards for the selection of health Measurement Instruments (COSMIN) team. Our study has been peer reviewed by a steering committee of 15 expert clinicians and academics and Nottingham University Hospital NHS foundation Trust's research committee. It is registered on the COSMIN database and will be published in a peer reviewed journal and on the NRC website on completion.

The modified Delphi study process will consist of a minimum of two phases with 2-4 rounds per phase.

E-Delphi software will be used to collect study data to decrease sample attrition and ensure anonymity and minimise power dynamics between participants.

The principal data holder will be the National Rehabilitation Centre as part of Nottingham University Hospitals Trust. The NRC will hold all rights for publication of the data, study protocol, full study report and anonymised participant level data. Authorship will be granted to aforementioned chief investigator and key contributors to this protocol, each of whom will also be involved in review of the final study results.

Full Methodology

Recruitment of the expert panel:

1. The NRC dataset steering committee or one of their nominees will recruit participants through purposive snowball sampling using standardised email invites
2. Each nominee will receive a document outlining the study background, aims, objectives, participant eligibility and methodology.
3. If participants agree to partake in the e-Delphi study they will contact the CI directly.
4. Upon receipt of a potential participant's expression of interest the CI will invite them to propose further study participants, outlining the specialist areas that still required on the expert panel. The participants will also be provided with a consent form and participant information sheet.
5. If nominees don't reply to invitations a follow-up email will be sent 10 days later. If there is no further communication, no further contact will be attempted.
6. If participants feel they meet the eligibility criteria, they must return a signed consent form to the CI as evidence of their intention to partake in the study. Participants are free to withdraw from the study at any time. No form of incentive will be provided.
7. The CI will countersign consent forms to confirm that study participants have signed and completed the form correctly. The participant is then assigned a study ID and provided with a copy of their countersigned consent form. At this point, the participant is asked to enter their professional experience and key demographic details into a JISC questionnaire. This information will be used to ensure that the expert panel is sufficiently diverse and represent the case-mix of patients being treated at the NRC.
8. The research team will confirm that the participant meets the eligibility criteria after reviewing the answers given in the JISC questionnaire.
9. Once a heterogenous panel of experts has been recruited or no further individuals are being nominated to be included in the expert panel, recruitment will close and the study will be formally launched.
10. At this point, all participant will be sent key documents and research papers, intended to inform their decision making during the Delphi process.
11. It is expected that the study will over-recruit by 20-30%, reaching a total of circa 50-60 individual participants. This allows for 2-3 experts in each field of practice.
12. Participants will be provided with a background document summarising the Rehabilitation Datasets being utilised internationally and key research papers relevant to the study.

    Phase 1:

    Exploring what information (data items) must be collected as part of the NRC's minimum dataset

    Round 1:
13. An initial list of proposed Core Data Items (outcome domains) agreed upon by the NRC dataset steering committee will be provided to the expert panel
14. These core data items (outcome domains) will include:

    i. Demographic information ii. Health indicators and associated outcome measures iii. Socio-economic data (healthcare costs, salary etc.) iv. Service delivery/care pathway variables (admission, transfer and discharge dates/locations etc.) v. Information associated with previous social function, employment and education and return to these activities following their injury/illness.

    vi. Injury/condition-specific data
15. Participants will priority rank each of the proposed data items based on the criteria outlined below.
16. Experts will also return a list of additional 'core' data items (outcome domains) they feel should be included in the National Rehabilitation Dataset by answering the question 'What additional data should be routinely collected for all rehabilitation patients in order to describe care and outcomes?'
17. At this time panel members will not be asked for matched outcome measures, but are encouraged to take note of these for later rounds and include them in comments. No limit will be placed on the number of data items proposed and participants will be encouraged to leave comments to express their opinion on any given item.

    Each data item will be ranked on a 9-point scale based on COMET initiative and OMERACT guidance as follows:

    (1-3) = 'Critical / Mandatory domains' (data that is considered essential for documentation and reporting the effectiveness and cost efficiency of the rehabilitation being provided)

    (4-6) = 'Important but not critical / important but optional domains' (data that improves the quality of data collected but is not critical to evaluating rehabilitation effectiveness and cost efficiency)

    (7-9) = 'Not that important / useful for research purposes' (optional data items that may supplement the core dataset for research purposes or specialist populations)

    Rounds 2-4:
18. All ranked data items will be anonymised and re-distributed to the expert panel. Each expert will evaluate their ranked responses before returning a final list to the Delphi coordinator. No limit will be placed on the required number of data items or health indicators that could be proposed.
19. The newly ranked list of data items will be re-distributed to the expert panel. Clearly outlining any uncertainties and disagreements to the expert panel for further consideration.
20. Any data item that has reached consensus of >70% after round 2 will be included in the final dataset. These core domains (data items) will then be excluded from subsequent rounds of voting.
21. If consensus is not met in round 2 then this round will be repeated until such a time that consensus is achieved prior to moving onto phase 2
22. If a consensus of >70% is not achieved in each of the core outcome domains after 4 round of voting, the highest-ranked responses with a consensus >60% will be accepted.
23. A written report summarising the proposed 'core' data items (outcome domains) will be distributed to the expert panel.
24. A video will be recorded by the study coordinator to present the consensus findings. Outlining the proposed 'core' data items and health indicators to be included in the NRC dataset, before outlining the next steps in the Delphi study.
25. Any ranked responses from phase 1 with 50-70% consensus as critical/mandatory that were not included in the final dataset will be included in the supplemental dataset alongside data items marked as 'important but not critical/optional domains' with a stable response rate.

    Phase 2: What tools should be used to evaluate the data items outlined in phase 1

    Round 1:
26. The expert panel will propose a list of outcome measure instruments to evaluate each of the proposed 'core' data items (inc. health indicators) identified in phase 1.
27. This list should be priority ranked based on the OMERACT and COSMIN checklists. Principally basing ranked choices on, (1) The appropriateness of the proposed outcome measure for the given population and (2) The quality of the outcome measure based on its reliability, validity, responsiveness to change and interpretability of the outcome data.
28. Where an outcome measure instrument is not required to measure fixed domains such as biological sex at birth or occupational status, the CI will include wording from the NHS data model/dictionary. Participants will be asked to comment on the domain wording.

    Ranked choices for each core data item will be ranks from 1-8 as follows:

    1-4 = Most appropriate outcome measure instrument / Domain 5-8 = Optional / supplemental outcome measure instrument / Domain that could be used for specific patient populations or for research purposes.

    Round 2-4:
29. The proposed outcome measures and their matched health indicators or data items will be anonymised and re-distributed to the expert panel, alongside a table outlining each outcome measure instrument's validity, reliability and responsiveness.
30. In round 2 participants will evaluate their ranked responses and return their final list.
31. A written report summarising the proposed 'core' data items and their associated outcome measure instruments, with any uncertainties / disagreements will be distributed to the expert panel.
32. Any outcome measure that has reached consensus of >70% will be included in the final dataset. The core domains (data items) these outcome measures assess will then be excluded from subsequent rounds of voting.
33. If consensus is not met in round 2 then this round will be repeated until such a time that consensus is achieved or 4 rounds are completed in phase 2. At this point the highest-ranked responses with a consensus >60% from each of the pre-identified categories will be accepted.
34. The finalised COS will be created and re-distributed to the panel for final approval alongside a short video presenting the consensus findings from phases 1 and 2 linking the study conclusions to International Classification of Disability and Health (ICF) core outcome sets and other relevant research.

Phase 3 (Optional):

If consensus was not achieved in phase 1 or 2 a nominal group technique will be used to reach consensus over the course of 1 working day.

During phase 3 the expert panel will discuss the supporting literature for each domain where uncertainty remains before voting on a final dataset.

If a consensus cannot be achieved, the meeting chair will have a deciding vote.

Data Analysis This study will use a mixed method approach of Quantitative and Qualitative analysis.

Quantitative analysis will include calculating the arithmetic mean and mode values before exploring standard deviations and interquartile ranges of the participant responses to represent the percentage agreement between participants' ratings (consensus). An outlier analysis will be completed to identify and exclude any results that could skew the interquartile range.

Qualitative analysis will include a thematic and content analysis of the statements each participant makes about a given topic or question using excel to aggregate and count similarly themed comments.

Thematic analysis will be coded as beliefs/opinions, differentiations, cause-effect relationships, examples, experiences, trends, no information, or misunderstandings.

Content analysis of participant's comments will be used to identify outcome measure instruments and other data items proposed by greater than one participant after each round. These will then be included into subsequent rounds of voting.

ELIGIBILITY:
Inclusion Criteria:

The panel will aim to include clinicians with a minimum of 5 years' experience from a variety of professional backgrounds within the following specialist areas:

* Neuro Rehab
* Trauma Rehab
* Community Rehab
* Outpatient Rehabilitation services
* Defence medical services
* Psychology services
* Amputee Rehab
* Speech and Language therapy
* Emergency department
* Critical Care
* Trauma and Orthopaedics
* Rehabilitation Medicine

It is expected that the expert panel will include:

* Medical Doctors
* Dietitians
* Physiotherapists
* Psychologists
* Prosthetists
* Occupational therapists
* Speech and Language therapists
* Data-base managers
* Researchers/Academics
* Commissioners
* Local service managers
* A department of work and pensions representative
* An epidemiologist/data-scientist with healthcare financial modelling experience

Exclusion Criteria:

Individuals will be excluded from the expert panel for any of the following reasons:

1. They do not have 5 years' experience in their specialist field
2. They do not have an understanding of various health indicators and the appropriate outcome measure instruments required to evaluate these health indicators.
3. They have no understanding of how demographic and socio-economic variables impact health outcomes
4. They have no understanding of how to evaluate clinical effectiveness and cost efficiency of inpatient rehabilitation services.
5. Their professional background is not represented in the above noted specialist areas

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The expert panel (study participants) will include clinicians, researchers and managers from a variety of fields. These experts will be purposefully selected based on their knowledge of how best to evaluate the clinical effectiveness and cost efficiency of inpatient rehabilitation services.
  This knowledge will include an understanding of which outcome measure instruments are most appropriate to monitor patients' health, social and economic outcomes and what demographic and socio-economic variables are important to record.
  The expert panel will have experience treating the cohort of patients that the National Rehabilitation Centre (NRC) will support or have experience developing trauma / rehabilitation registries.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2025-01 (Estimated); Primary Completion 2025-06 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
To develop a Core Outcome Set (COS) for rehabilitation to be used as the foundation of the National Rehabilitation Centre Dataset. | From enrolment to conclusion of the stufy (6 months)
  The core outcome set (Primary outcome) will include core data Items centered on 6 key themes:
  1. Demographic variables
  2. Health indicators and associated outcome measures
  3. Socio-economic variables (healthcare costs, salary etc.)
  4. Service delivery/care pathway variables (admission, transfer and discharge dates/locations etc.)
  5. Information associated with previous social function, employment and education and return to these activities following their injury/illness.
  6. Injury/condition-specific data
  Each data item will include details regarding how this item will be measured

OTHER OUTCOMES:
To develop a Core Outcome Set (COS) for rehabilitation to be used as the foundation of the National Rehabilitation Centre Dataset. | From enrolment to conclusion of the study (6 months)
  The core outcome set (Primary outcome) will include core data Items centred on 6 key themes:
  1. Demographic variables
  2. Health indicators and associated outcome measures
  3. Socio-economic variables (healthcare costs, salary etc.)
  4. Service delivery/care pathway variables (admission, transfer and discharge dates/locations etc.)
  5. Information associated with previous social function, employment and education and return to these activities following their injury/illness.
  6. Injury/condition-specific data

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Corbett, MSc, Principal Investigator — Research at the National Rehabilitation Centre (part of Nottingham University Hospital NHS Trust)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Young AM, Chung H, Chaplain A, Lowe JR; STARS Rehabilitation Dataset Development Group; Wallace SJ. Development of a minimum dataset for subacute rehabilitation: a three-round e-Delphi consensus study. BMJ Open. 2022 Mar 25;12(3):e058725. doi: 10.1136/bmjopen-2021-058725. PMID 35338067
- [Background] Hernandez-Segura N, Marcos-Delgado A, Pinto-Carral A, Fernandez-Villa T, Molina AJ. Health-Related Quality of Life (HRQOL) Instruments and Mobility: A Systematic Review. Int J Environ Res Public Health. 2022 Dec 8;19(24):16493. doi: 10.3390/ijerph192416493. PMID 36554369
- [Background] Herdman M, Gudex C, Lloyd A, Janssen M, Kind P, Parkin D, Bonsel G, Badia X. Development and preliminary testing of the new five-level version of EQ-5D (EQ-5D-5L). Qual Life Res. 2011 Dec;20(10):1727-36. doi: 10.1007/s11136-011-9903-x. Epub 2011 Apr 9. PMID 21479777
- [Background] Cieza A, Kirchberger I, Biering-Sorensen F, Baumberger M, Charlifue S, Post MW, Campbell R, Kovindha A, Ring H, Sinnott A, Kostanjsek N, Stucki G. ICF Core Sets for individuals with spinal cord injury in the long-term context. Spinal Cord. 2010 Apr;48(4):305-12. doi: 10.1038/sc.2009.183. Epub 2010 Jan 12. PMID 20065984
- [Background] Fresk M, Grooten WJA, Brodin N, Backlund LG, Arrelov B, Skaner Y, Kiessling A. Mapping information regarding the work-related disability of depression and long-term musculoskeletal pain to the International Classification of Functioning, Disability and Health and ICF Core Sets. Front Rehabil Sci. 2023 May 2;4:1159208. doi: 10.3389/fresc.2023.1159208. eCollection 2023. PMID 37200737
- [Background] Cieza A, Stucki G, Weigl M, Kullmann L, Stoll T, Kamen L, Kostanjsek N, Walsh N. ICF Core Sets for chronic widespread pain. J Rehabil Med. 2004 Jul;(44 Suppl):63-8. doi: 10.1080/16501960410016046. PMID 15370750
- [Background] Oral A, Kiekens C, DE Vriendt P, Satink T, VAN DE Velde D, Grazio S, Moslavac S, Schnurrer-Luke-Vrbanic T, Vlak T, Kontaxakis A, Rapidi CA, Pyrgeli M, Stavrianou A, Kujawa J, Tederko P, Kucukdeveci AA, Sezgin M, Zampolini M, Stucki G, Selb M. Development of simple descriptions of the ICF Generic-30 Set in different languages: laying the foundation for an ICF-based clinical tool for Europe. Eur J Phys Rehabil Med. 2023 Jun;59(3):271-283. doi: 10.23736/S1973-9087.23.07932-7. Epub 2023 Apr 21. PMID 37083101
- [Background] Dworkin RH, Turk DC, Farrar JT, Haythornthwaite JA, Jensen MP, Katz NP, Kerns RD, Stucki G, Allen RR, Bellamy N, Carr DB, Chandler J, Cowan P, Dionne R, Galer BS, Hertz S, Jadad AR, Kramer LD, Manning DC, Martin S, McCormick CG, McDermott MP, McGrath P, Quessy S, Rappaport BA, Robbins W, Robinson JP, Rothman M, Royal MA, Simon L, Stauffer JW, Stein W, Tollett J, Wernicke J, Witter J; IMMPACT. Core outcome measures for chronic pain clinical trials: IMMPACT recommendations. Pain. 2005 Jan;113(1-2):9-19. doi: 10.1016/j.pain.2004.09.012. No abstract available. PMID 15621359
- [Background] Beiderbeck D, Frevel N, von der Gracht HA, Schmidt SL, Schweitzer VM. Preparing, conducting, and analyzing Delphi surveys: Cross-disciplinary practices, new directions, and advancements. MethodsX. 2021 May 28;8:101401. doi: 10.1016/j.mex.2021.101401. eCollection 2021. PMID 34430297
- [Background] Kirkham JJ, Gorst S, Altman DG, Blazeby JM, Clarke M, Devane D, Gargon E, Moher D, Schmitt J, Tugwell P, Tunis S, Williamson PR. Core Outcome Set-STAndards for Reporting: The COS-STAR Statement. PLoS Med. 2016 Oct 18;13(10):e1002148. doi: 10.1371/journal.pmed.1002148. eCollection 2016 Oct. PMID 27755541
- [Background] Kirkham JJ, Davis K, Altman DG, Blazeby JM, Clarke M, Tunis S, Williamson PR. Core Outcome Set-STAndards for Development: The COS-STAD recommendations. PLoS Med. 2017 Nov 16;14(11):e1002447. doi: 10.1371/journal.pmed.1002447. eCollection 2017 Nov. PMID 29145404
- [Background] Schmitt J, Apfelbacher C, Spuls PI, Thomas KS, Simpson EL, Furue M, Chalmers J, Williams HC. The Harmonizing Outcome Measures for Eczema (HOME) roadmap: a methodological framework to develop core sets of outcome measurements in dermatology. J Invest Dermatol. 2015 Jan;135(1):24-30. doi: 10.1038/jid.2014.320. Epub 2014 Sep 4. PMID 25186228
- [Background] Boers M, Kirwan JR, Wells G, Beaton D, Gossec L, d'Agostino MA, Conaghan PG, Bingham CO 3rd, Brooks P, Landewe R, March L, Simon LS, Singh JA, Strand V, Tugwell P. Developing core outcome measurement sets for clinical trials: OMERACT filter 2.0. J Clin Epidemiol. 2014 Jul;67(7):745-53. doi: 10.1016/j.jclinepi.2013.11.013. Epub 2014 Feb 28. PMID 24582946
- [Background] Nasa P, Jain R, Juneja D. Delphi methodology in healthcare research: How to decide its appropriateness. World J Methodol. 2021 Jul 20;11(4):116-129. doi: 10.5662/wjm.v11.i4.116. eCollection 2021 Jul 20. PMID 34322364
- [Background] Gattrell WT, Logullo P, van Zuuren EJ, Price A, Hughes EL, Blazey P, Winchester CC, Tovey D, Goldman K, Hungin AP, Harrison N. ACCORD (ACcurate COnsensus Reporting Document): A reporting guideline for consensus methods in biomedicine developed via a modified Delphi. PLoS Med. 2024 Jan 23;21(1):e1004326. doi: 10.1371/journal.pmed.1004326. eCollection 2024 Jan. PMID 38261576
- [Background] NCASRI Project team, Lead: Turner-Stokes L., 'Specialist Rehabilitation following major Injury (NCASRI) Final Audit report'.
- [Background] Prinsen CA, Vohra S, Rose MR, Boers M, Tugwell P, Clarke M, Williamson PR, Terwee CB. How to select outcome measurement instruments for outcomes included in a "Core Outcome Set" - a practical guideline. Trials. 2016 Sep 13;17(1):449. doi: 10.1186/s13063-016-1555-2. PMID 27618914
- [Background] Williamson PR, Altman DG, Bagley H, Barnes KL, Blazeby JM, Brookes ST, Clarke M, Gargon E, Gorst S, Harman N, Kirkham JJ, McNair A, Prinsen CAC, Schmitt J, Terwee CB, Young B. The COMET Handbook: version 1.0. Trials. 2017 Jun 20;18(Suppl 3):280. doi: 10.1186/s13063-017-1978-4. PMID 28681707